CLINICAL TRIAL: NCT07323602
Title: Prediction of Deep Brain Stimulation (DBS) Efficacy in Patients With Dystonia Based on Preoperative Wearable Gait Analysis: A Prospective Observational Study
Brief Title: Predicting DBS Outcomes in Dystonia Using Wearable Gait Sensors
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Collaborators: Suzhou Sceneray Medical Co. , Ltd (Industry); Beijing Pins Medical Co., Ltd (Industry); Medtronic (Industry)
Responsible Party: Principal Investigator, LI DIANYOU, Doctor, Ruijin Hospital
Other Study IDs: DYSGAITpredictDBS
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Dystonia
Keywords: dystonia; deep brain stimulation; wearable Gait Analysis
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Wearable Gait Sensor Analysis — Patients will wear inertial measurement units (IMUs) on [specify body parts, e.g., lower back, ankles] to record gait data during standardized walking tasks before surgery.

SUMMARY:
This study aims to investigate whether preoperative gait characteristics, measured by wearable sensors, can predict the clinical outcomes of Deep Brain Stimulation (DBS) in patients with dystonia. Participants scheduled for DBS surgery will undergo gait analysis using wearable sensors before the procedure. Clinical assessments, including the Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) and the SF-36 Health Survey, will be conducted preoperatively and postoperatively to evaluate surgical efficacy and quality of life. The study seeks to identify gait biomarkers that correlate with optimal DBS response.

DETAILED DESCRIPTION:
This study aims to investigate whether preoperative gait characteristics, measured by wearable sensors, can predict the clinical outcomes of Deep Brain Stimulation (DBS) in patients with dystonia. Participants scheduled for DBS surgery will undergo gait analysis using wearable sensors before the procedure. Clinical assessments, including the Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) and the SF-36 Health Survey, will be conducted preoperatively and postoperatively to evaluate surgical efficacy and quality of life. The study seeks to identify gait biomarkers that correlate with optimal DBS response.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with primary or isolated dystonia.
* Scheduled to undergo bilateral Deep Brain Stimulation (DBS) surgery.
* Able to walk independently or with assistance (sufficient to perform gait analysis).
* Willing to participate and sign informed consent.

Exclusion Criteria:

* History of other neurological disorders affecting gait (e.g., stroke, severe neuropathy).
* Significant orthopedic issues preventing gait assessment.
* Cognitive impairment preventing cooperation with study procedures.
* Previous functional neurosurgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients clinically diagnosed with isolated dystonia who are candidates for Deep Brain Stimulation (DBS) surgery at Ruijin Hospital. These participants have motor symptoms that are refractory to optimal medical therapy and are scheduled for elective surgical intervention.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between Baseline Gait Features and BFMDRS Improvement | Through study completion, up to 6 months

SECONDARY OUTCOMES:
Change in Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) Score | Baseline (pre-operative) and 6 months post-operative
Change in SF-36 Quality of Life Score | Baseline (pre-operative) and 6 months post-operative
Gait Characteristics (Spatio-temporal parameters) | Baseline (pre-operative)

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China